CLINICAL TRIAL: NCT05373446
Title: Evaluation of SSD8432 in Combination With Ritonavir in Asymptomatic Infections or Mild/Common Randomized, Double-blind, Safety Study of Efficacy and Safety in Adult Subjects With COVID-19 Placebo-Controlled, Phase II Clinical Study
Brief Title: Evaluation of SSD8432 and Ritonavir in Adult Subjects With COVID-19 Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B02B11101-201
Record Dates: First submitted 2022-05-12; First posted 2022-05-13 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SIM0417; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSD8432 300mg (Experimental): SSD8432 300mg in combination with ritonavir 100mg
  Interventions: Drug: SSD8432 300mg
- SSD8432 750mg (Experimental): SSD8432 750mg in combination with ritonavir 100mg
  Interventions: Drug: SSD8432 750mg
- SSD8432 placebo (Placebo Comparator): SSD8432 placebo in combination with ritonavir placebo
  Interventions: Drug: SSD8432Placebo

INTERVENTIONS:
Drug: SSD8432 300mg — SSD8432 300mg in combination with ritonavir 100mg, day1--day5,BID
  Other Names: ritonavir 100mg
  Arms: SSD8432 300mg
Drug: SSD8432 750mg — SSD8432 750mg in combination with ritonavir 100mg, day1--day5,BID
  Other Names: ritonavir 100mg
  Arms: SSD8432 750mg
Drug: SSD8432Placebo — SSD8432Placebo in combination with ritonavir placebo,day1--day5,BID
  Other Names: ritonavir placebo
  Arms: SSD8432 placebo

SUMMARY:
This is a Randomized, double-blind, Placebo-Controlled, Phase II Clinical Study to evaluate SSD8432 in combination with Ritonavir in asymptomatic infections or mild/common safety study of efficacy and safety in adult subjects with COVID-19.

DETAILED DESCRIPTION:
This is a Randomized, double-blind, Placebo-Controlled, Phase II Clinical Study to evaluate SSD8432 in combination with Ritonavir in asymptomatic infections or mild/common safety study of efficacy and safety in adult subjects with COVID-19.

This study planned to enroll 72 subjects, randomly divided into low-dose group, high-dose group and placebo group according to 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤80 years old, male or female.
2. Asymptomatic infection,mild or common type of COVID-19.
3. Initial positive test of SARS-CoV-2 within 5 days of randomization.
4. Initial onset of COVID-19 signs/symptoms within 3 days of randomization.

Exclusion Criteria:

1. Transnasal high-flow oxygen therapy or non-invasive ventilation, invasive mechanical ventilation, or ECMO is required or anticipated to be urgently required.
2. Prior to current disease episode, any confirmed SARS-CoV-2 infection.
3. Known medical history of active liver disease (other than nonalcoholic hepatic steatosis).
4. Receiving dialysis or have known moderate to severe renal impairment.
5. Known human immunodeficiency virus (HIV) infection.
6. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
7. Oxygen saturation of ≤ 93% on room air obtained at rest within 24 hours prior to randomization..
8. Treatment with antivirals against SARS-CoV-2 within 14 days.
9. Current or expected use of any medications or substances that are highly dependent on CYP3A4 for clearance.
10. Concomitant use of any medications or substances that are strong inducers of CYP3A4 are prohibited within 28 days.
11. Has received or is expected to receive COVID-19 monoclonal antibody, convalescent COVID-19 plasma or other prohibited concomitant medication.
12. Females who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to first nucleic acid turning negative | Baseline through Day28
  The time from the first administration to the first nucleic acid turning negative

SECONDARY OUTCOMES:
viral load | Baseline through Day28
  Changes of viral load compared to the baseline
adverse events | Baseline through Day28
  Frequency of TEAE
Time to Sustained Alleviation | baseline through Day28
  Time to Sustained Alleviation of Targeted COVID-19 Signs/symptoms
Resting oxygen saturation | Day1 and Day5
  Proportion of subjects with resting oxygen saturation ≥ 95%
Proportion of participants progressing to a worsening status(higher score) | Baseline through Day28
  WHO clinical progression scale(0 to 10)
Maximum plasma concentration(Cmax) | Baseline through Day5
  Plasma concentration of SSD8432

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Yang, doctor, Study Director — Jiangsu Xiansheng Pharmaceutical Co.,

IPD SHARING:
Plan to Share IPD: No